CLINICAL TRIAL: NCT03875079
Title: An Open-Label, Multicenter, Phase Ib Study to Evaluate Safety and Therapeutic Activity of RO6874281, an Immunocytokine, Consisting of Interleukin-2 Variant (IL-2v) Targeting Fibroblast Activation Protein-Α (FAP), in Combination with Pembrolizumab (Anti-PD-1), in Participants with Advanced or Metastatic Melanoma
Brief Title: A Study to Evaluate Safety and Therapeutic Activity of RO6874281 in Combination with Pembrolizumab, in Participants with Advanced or Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP41054; 2018-003872-11 (EudraCT Number)
Record Dates: First submitted 2019-03-13; First posted 2019-03-14 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part I Safety Run in: RO6874281 + Pembrolizumab (Experimental): Cohort 1.1 (CPI naive and experienced melanoma participants):
  Participants will receive RO6874281 in combination with Pembrolizumab every 3 weeks (Q3W) and will be observed for 2 cycles (ie: 6 weeks) in order to confirm the safety of the proposed dose and schedule that will be used in Part II of this study.
  Cohort 1.2 (CPI experienced melanoma participants only):
  Participants will receive RO6874281 in combination with Pembrolizumab via an induction and maintenance schedule for RO6874281: QW three times (D1, D8, D15) followed by Q3W dosing (D22 and subsequent). Pembrolizumab is to be administered Q3W, starting on Day 1. Participants will be observed for 2 pembrolizumab cycles (ie: 6 weeks) in order to confirm the safety of the proposed dose and schedule that will be used in Part III of this study.
  Interventions: Drug: RO6874281; Drug: Pembrolizumab
- Part II Expansion: RO6874281 + Pembrolizumab (Experimental): Part II will start once all participants in Part I Cohort 1.1 have completed the observation period. Approximately 34 participants will receive RO6874281 in combination with Pembrolizumab every 3 weeks (Q3W) and will be observed for 2 cycles (ie: 6 weeks).
  Interventions: Drug: RO6874281; Drug: Pembrolizumab
- Part III Expansion: RO6874281 + Pembrolizumab (Experimental): Part III will start once all participants in Part I Cohorts 1.1 and 1.2 have completed the observation period. Approximately 80 participants will be randomised to receive RO6874281 in combination with Pembrolizumab in either a Q3W or QW/Q3W schedule.
  Interventions: Drug: RO6874281; Drug: Pembrolizumab

INTERVENTIONS:
Drug: RO6874281 — Part I Safety Run in:
  Cohort 1.1: RO6874281 will be administered by intravenous (IV) infusion; 10 mg (Q3W) every 3 weeks and will be observed over 2 administration cycles (i.e. 6 weeks) in order to confirm the safety of the proposed dose and schedule that will be used in Part II of this study.
  Cohort 1.2: RO6874281 will be administered by IV infusion via an induction and maintenance phase; 10 mg (QW) every week for 3 weeks followed by 10 mg (Q3W) every 3 weeks and will be observed over 2 administration cycles (6 weeks) to confirm safety of the proposed dose and schedule to be used in Part III of this study.
  Part II Expansion: RO6874281 will be administered by IV infusion; 10 mg (Q3W) every 3 weeks (or lower dose level depending on Part I Cohort 1.1 outcome).
  Part III Expansion: RO6874281 will be administered by IV infusion; 10 mg (QW) every week or 10mg (Q3W) every 3 weeks (or lower dose level depending on Part I Cohorts 1.1 and 1.2 outcomes) in either a Q3W or QW/Q3W schedule.
  Other Names: simlukafusp alfa
Drug: Pembrolizumab — Part I Safety Run in (Cohorts 1.1 and 1.2): Pembrolizumab will be administered by IV; 200 mg Q3W and will be observed over 2 administration cycles (i.e. 6 weeks).
  Part II Expansion: Pembrolizumab will be administered by IV; 200 mg Q3W (or lower dose level depending on Part I Cohort 1.1 outcome)
  Part III Expansion: Pembrolizumab will be administered by IV; 200 mg Q3W (or lower dose level depending on Part I Cohorts 1.1 and 1.2 outcomes)

SUMMARY:
This is an open-label, multicenter, Phase Ib study to evaluate the safety and therapeutic activity of RO6874281 in combination with pembrolizumab. The study will consist of 3 parts: a safety run-in (Part I: Cohorts 1.1. and 1.2) and two expansion parts (Parts II and III). Part II will start once all participants in Cohort 1.1 have completed the observation period. Part III will start once all participants in Cohorts 1.1 and 1.2 have completed the observation period.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed unresectable stage III or stage IV cutaneous or mucosal melanoma (AJCC v8.0).
2. Participants need to have known BRAF status.
3. CPI naïve melanoma population: Participants with unresectable stage III or stage IV cutaneous or mucosal melanoma who have not received prior treatment for advanced disease. BRAF mutation-positive patients are eligible without prior treatment or after failure of BRAF directed inhibitor therapy.
4. CPI experienced melanoma population: Participants with unresectable stage III or stage IV cutaneous melanoma. Participants must have progressed during or after treatment with anti PD-1 antibody therapy, either as monotherapy or in combination with other agent(s).
5. Participants should have adequate cardiovascular, hematological, liver, and renal function.
6. Participants with unilateral pleural effusion are eligible if they fulfill both of the following: NYHA Class 1; Forced expiratory volume 1 (FEV1) >70% and forced vital capacity (FVC) >70% of predicted value; participants with lung metastases should present with DLCO >60% of predicted value.

Exclusion criteria:

Medical Conditions

1. Rapid disease progression or suspected hyperprogression (as determined by the Investigator) or threat to vital organs or critical anatomical sites requiring urgent alternative medical intervention.
2. Known active CNS metastases and/or carcinomatous meningitis/leptomeningeal disease:

   Participants with previously treated brain metastases may participate.
3. History of treated asymptomatic CNS metastases.
4. An active second malignancy (exceptions are non-melanoma skin cancer, cervical carcinoma in situ, or prostate carcinoma that is in remission under androgen deprivation therapy for ≥ 2 years, or participants who have a history of malignancy and have been treated with curative intent and the participant is expected to be cured as per Investigator's assessment).
5. Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results, and known autoimmune diseases or other disease with ongoing fibrosis (such as scleroderma, pulmonary fibrosis. and emphysema).
6. Episode of significant cardiovascular/cerebrovascular acute disease within 6 months before study treatment administration.
7. Active or uncontrolled infections, including latent tuberculosis.
8. Known HIV infection.
9. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
10. Severe infection within 4 weeks before study treatment administration, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia.
11. History of chronic liver disease or evidence of hepatic cirrhosis.
12. Dementia or altered mental status that would prohibit informed consent.
13. History of autoimmune disease.
14. Adverse events related to any previous radiotherapy, chemotherapy, targeted therapy, CPI therapy or surgical procedure that have not resolved to Grade =< 1, except alopecia (any grade) and Grade 2 peripheral neuropathy.
15. History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan.
16. Bilateral pleural effusion.
17. Severe dyspnea at rest or requiring supplementary oxygen therapy.
18. Concurrent therapy with any other investigational drug (defined as a treatment for which there is currently no regulatory authority approved indication).
19. Immunomodulating agents: Last dose with any of the following agents, for example, etanercept, infliximab, tacrolimus, cyclosporine, mycophenolic acid, alefacept, or efalizumab (or similar agents) < 28 days before study treatment administration. Regular immunosuppressive therapy (i.e., for organ transplantation, chronic rheumatologic disease)
20. Treatment with systemic immunosuppressive medications including, but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF agents within 2 weeks prior to Cycle 1 Day 1.
21. Radiotherapy within the last 4 weeks before start of study treatment administration, with the exception of limited field palliative radiotherapy.
22. Administration of a live, attenuated vaccine within 4 weeks before Cycle 1 Day 1.
23. Major surgery or significant traumatic injury < 28 days before study treatment administration (excluding fine needle biopsies) or anticipation of the need for major surgery during study treatment.
24. Known hypersensitivity to any of the components of the RO6874281 drug product or pembrolizumab drug product, including but not limited to hypersensitivity to Chinese Hamster Ovary cell products or other recombinant human or humanized antibodies.
25. No prior cytotoxic therapy for unresectable stage III or stage IV disease is permitted.
26. Toxicity from prior anti-PD-1 antibody therapy (including adjuvant treatment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with adverse events | Baseline to end of study (approximately 24 months)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Time from first occurrence of a documented objective response until the time of documented disease progression or death from any cause during treatment (whichever occurs first) until the end of study (approximately 24 months)
Complete Response Rate (CRR) | Baseline to end of study (approximately 24 months)
Disease Control Rate (DCR) | Baseline to end of study (approximately 24 months)
Duration of Response | Time from first occurrence of a documented objective response until the time of documented disease progression or death from any cause during treatment (whichever occurs first) until the end of study (approximately 24 months)
Progression Free Survival (PFS) | Time from study treatment initiation to the first occurrence of documented disease progression (based on Investigator's assessment) or death from any cause during treatment (whichever occurs first) until the end of study (approximately 24 months)
Baseline PD-L1 | Baseline to end of study (approximately 24 months)
Fibroblast Activation Protein-a (FAP) | Baseline to end of study (approximately 24 months)
Change from baseline in density (cell/mm2) of immune cells including CD8+, FOXP3, and PD-L1 | Baseline to end of study (approximately 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- United States (4):
  - Yale University, New Haven, Connecticut
  - University of Iowa, Iowa City, Iowa
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
- Australia (2):
  - Melanoma Institute Australia, North Sydney, New South Wales
  - Peter Maccallum Cancer Institute; Clinical Trial Unit, Melbourne, Victoria
- Belgium (2):
  - UZ Antwerpen, Edegem
  - UZ Leuven Gasthuisberg, Leuven
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- France (4):
  - Hopital Claude Huriez; Sce Dermatologie, Lille
  - Hôpital de la Timone; Dermatologie, Marseille
  - Centre Eugene Marquis; Service d'oncologie, Rennes
  - Institut Gustave Roussy; Dermatologie, Villejuif
- Russia (4):
  - Main Military Clinical Hospital named after N.N. Burdenko, Moscow, Moscow Oblast
  - Russian Oncology Research Center n.a. N.N. Blokhin, Moscow
  - P.A. Gertsen Cancer Research Inst. ; Chemotherapy Dept, Moscow
  - FBI "Scientific Research Institute of Oncology n. a. N. N. Petrov", Saint Petersburg
- Spain (5):
  - Hospital Universitari Vall d'Hebron; Oncology, Barcelona, BARCELONA
  - Hospital Clínic i Provincial; Servicio de Oncología, Barcelona, BARCELONA
  - Clinica Universidad de Navarra Madrid; Servicio de Oncología, Madrid, Madrid
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid, Madrid
  - Clinica Universitaria de Navarra; Servicio de Oncologia, Pamplona, Navarre

IPD SHARING:
Plan to Share IPD: No
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing